CLINICAL TRIAL: NCT02457728
Title: Mesh Fixation and Closure of Peritoneum Following Laparoscopic Hernia Repair Using N-butyl Cyanoacrylate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St John of God Hospital, Vienna (Other)
Responsible Party: Principal Investigator, Bernhard Dauser, MD, MD, St John of God Hospital, Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: StJohn
Record Dates: First submitted 2015-05-17; First posted 2015-05-29 (Estimated); Results first posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-10

CONDITIONS: Hernia, Inguinal
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inguinal herniation (Experimental): In patients with bilateral herniations it should be explored if one glue device (LiquiBandFix8) for mesh fixation and closure of peritoneum is sufficient.
  Interventions: Device: LiquiBandFix8

INTERVENTIONS:
Device: LiquiBandFix8 — Using LiquiBandFix8 for mesh fixation and peritoneal closure following TAPP repair.

SUMMARY:
Fixation of mesh and peritoneal closure during TAPP repair using n-butyl cyanoacrylate.

DETAILED DESCRIPTION:
During transabdominal pre peritoneal (TAPP) hernia repair a mesh should be fixed at four pre-determined points. Number of attempts to fix the mesh with a novel non-penetrating fixation device (LiquiBandFix8) will be recorded. This novel device uses n-butyl cyanoacrylate and a defined amount of glue can be delivered with this 5mm laparoscopic instrument (liquid anchors).

In addition, closure of peritoneum should be accomplished using this device.

ELIGIBILITY:
Inclusion Criteria:

* Inguinal hernia,
* femoral hernia

Exclusion Criteria:

* pregnancy,
* not able to understand patient information

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard DAUSER, MD, Principal Investigator — St John of God Hospital, Vienna
Locations (1):
- St John of God Hospital, Graz, Styria, Austria

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Inguinal Herniation
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Inguinal Herniation: In patients with bilateral herniations it should be explored if one glue device (LiquiBandFix8) for mesh fixation and closure of peritoneum is sufficient.
  LiquiBandFix8: Using LiquiBandFix8 for mesh fixation and peritoneal closure following TransAbdominalPrePeritoneal (TAPP) repair.
Arm/Group | Inguinal Herniation
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 30
Region of Enrollment [Number; unit: participants]
  Austria | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Safe Fixation of Mesh and Closure of Peritoneum by Clinical Investigation During Hospital Stay and Telephone Interview at Six Weeks Postoperatively.
Description: Clinical examination during hospital stay to rule out any bowel obstruction due to insufficient closure of peritoneum. Telephone interview at six weeks postoperatively to record any adverse events in the early postoperative period such as recurrent hernia, pain or bowel obstruction.
Time Frame: During hospitalization and 6 weeks after surgery.
Measure: Number; unit: participants
Groups:
- Single-port TAPP Repair: LiquiBandFix8 for mesh fixation and peritoneal closure following TAPP repair using a single-port approach.
Arm/Group | Single-port TAPP Repair
Number analyzed (Participants) | 34
participants | 6

ADVERSE EVENTS:
Time Frame: 2 months
Groups:
- TAPP Repair: LiquiBandFix8 for mesh fixation and peritoneal closure following TAPP repair.
Arm/Group | TAPP Repair
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 6/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAPP Repair (N=34)
clogging of device (Surgical and medical procedures) | 5 (5) — Malfunction of device by clogging of the tip was recorded.
Persistent pain (Injury, poisoning and procedural complications) | 1 (1) — Persistent pain in the groin following TAPP repair

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No